CLINICAL TRIAL: NCT03966872
Title: Comparative Effectiveness of Integrated Illness Management and Recovery Versus the Chronic Disease Self-Management Program
Brief Title: Comparative Effectiveness of IIMR Versus CDSMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Sarah Pratt, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: D19103 31245
Record Dates: First submitted 2019-05-01; First posted 2019-05-29 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Mental Illness; Chronic Disease
Keywords: integrated health; mental health; illness management; cardiovascular disease; physical health
MeSH Terms: conditions — Mental Disorders; Chronic Disease; Psychological Well-Being; Cardiovascular Diseases | interventions — Salvage Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Illness Management and Recovery (I-IMR): (Experimental): Participants assigned to I-IMR will receive 2 individual sessions to discuss principles of recovery and set personally meaningful goals, with the remainder of the 14 I-IMR sessions delivered in groups of 8-10 (to enable individual tailoring)
  Interventions: Behavioral: Integrated Illness Management and Recovery
- Stanford Chronic Disease Self-Management Program (CDSMP): (Experimental): Participants randomly assigned get a 6-session group-based educational program co-delivered by two peers (lay people who have successfully managed a chronic illness) or a peer and a professional
  Interventions: Behavioral: Chronic Disease Self-Management Program

INTERVENTIONS:
Behavioral: Integrated Illness Management and Recovery — Education and skills training groups on illness management of chronic medical and psychiatric illness.
  Arms: Integrated Illness Management and Recovery (I-IMR):
Behavioral: Chronic Disease Self-Management Program — Education and skills training groups on illness management of chronic conditions
  Arms: Stanford Chronic Disease Self-Management Program (CDSMP):

SUMMARY:
The study will enroll 600 people with serious mental illness who receive services at Centerstone in KY or TN and will compare two different evidence-based self-management interventions: Integrated Illness Management and Recovery (I-IMR), a program developed by the study team at Dartmouth that trains people with serious mental illness on physical and mental health self-management, and the Stanford Chronic Disease Self-Management Program (CDSMP), a program largely focused on physical health self-management that has been used widely in the general population.

DETAILED DESCRIPTION:
The proposed study will be the first to compare two commonly used but substantially different, evidence-based self-management interventions. Integrated Illness Management and Recovery (I-IMR), is an individually-tailored, 16-session, integrated program combining both physical and mental health self-management specifically developed for people with SMI. In contrast, the Stanford Chronic Disease Self-Management Program (CDSMP) is a group-based, 6-session, chronic disease self-management program largely focused on physical health self-management alone. I-IMR is delivered by community mental health providers or by community outreach workers, while CDSMP is co-delivered by two peers or by a health professional and a peer. Both programs have been widely recommended, disseminated, and used. The proposed parent study will randomize people with serious mental illness to I-IMR (n=300) and CDSMP (n=300).

ELIGIBILITY:
Inclusion Criteria:

* Serious Mental Illness (diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or chronic depression with moderate impairment in functioning) receiving services at Centerstone(KY and TN)
* Diagnosis of a chronic medical condition increasing risk of early mortality from cardiovascular or respiratory disease (e.g., diabetes, hyperlipidemia, hypertension, COPD, heart failure, tobacco dependence, obesity), and at least 1 ER visit or hospitalization within the past year or judgment by the treatment team of substantial need for illness self-management training.

Exclusion Criteria:

* Consumers who do not speak English
* Consumers with either no, or a well-controlled medical condition will not be included
* Individuals residing in a nursing home or other institution
* Evidence of significant cognitive impairment as indicated by a Mini Mental Status Examination score <24, will be excluded

Eligibility for the COVID -related substudy is dependent on enrollment and participation in the parent project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knowledge and skills in illness self-management using the Illness Management and Recovery Scale | Change from Baseline to 12 months
  Change in knowledge and skills for illness self-management. Range of scores from 15-75 with higher scores meaning better illness self-management.
Change in Patient Activation on the Patient Activation Measure (PAM) | Change from Baseline to 12 months
  Change in Patient Activation (engagement in health care). Maximum score of 100, higher scores meaning greater activation.
Change in Acute Hospital Events from Electronic Medical Record Review. | Change from Baseline to 12 months
  Change in the number of acute hospital events. At each assessment a combination of participant report and verified information from mental health clinics will be used to validate the number acute hospital events.
Knowledge and Behaviors for Preventing Catching and Spreading COVID-19 Scale | Change from Baseline to 12 weeks
  Change in score on this measure, which was developed as part of the study plan because no suitable scale existed to assess knowledge and safety behaviors for COVID-19. Scores range from 0-100%, with higher scores indicating greater knowledge and enactment of safety behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pratt, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (2):
- United States (2):
  - Seven Counties Services, Louisville, Kentucky
  - Centerstone, Nashville, Tennessee